CLINICAL TRIAL: NCT00922038
Title: Encouraging Safe Sexual Practices Among Youth Using Cash Rewards: A Randomized Trial in the Kilombero/Ulanga Districts, Tanzania
Brief Title: Rewarding Sexually Transmitted Infection (STI) Prevention and Control in Tanzania
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: World Bank (Other); Health Effects Institute (Other); William and Flora Hewlett Foundation (Other); Population Health Research Institute (Other); University of California, San Francisco (Other); RTI International (Other)
Responsible Party: William H. Dow, Associate Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 025202
Record Dates: First submitted 2009-06-12; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High reward (Experimental)
  Interventions: Behavioral: Cash reward
- Low reward (Experimental)
  Interventions: Behavioral: Cash reward
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Cash reward — Enrollees testing negative for treatable sexually transmitted infections will receive cash rewards.
  Arms: High reward; Low reward

SUMMARY:
This project evaluates the effect of a combined economic and psycho-social intervention to reduce risky sexual activity and its consequences. The main hypothesis to be tested is that risky sexual activity and resulting sexually transmitted infections (STIs) can be reduced through an intervention of counseling, regular STI testing, and positive reinforcement using cash rewards. The intervention is being implemented in a population of young people in rural Tanzania where more conventional behavioral change interventions have had limited effect in battling a generalized HIV epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Plan to live in study area for next 12 months

Exclusion Criteria:

* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2411 (Actual)
Dates: Start 2009-02

PRIMARY OUTCOMES:
Prevalence of sexually transmitted infections measured in laboratory testing (Chlamydia, Gonorrhea, Syphilis, Trichomonas, Mycoplasma genitalium, HSV-2, HIV) | 4, 8, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William H Dow, PhD, Principal Investigator — University of California, Berkeley

REFERENCES:
- [Derived] de Walque D, Dow WH, Nathan R, Abdul R, Abilahi F, Gong E, Isdahl Z, Jamison J, Jullu B, Krishnan S, Majura A, Miguel E, Moncada J, Mtenga S, Mwanyangala MA, Packel L, Schachter J, Shirima K, Medlin CA. Incentivising safe sex: a randomised trial of conditional cash transfers for HIV and sexually transmitted infection prevention in rural Tanzania. BMJ Open. 2012 Feb 8;2(1):e000747. doi: 10.1136/bmjopen-2011-000747. Print 2012. PMID 22318666